CLINICAL TRIAL: NCT02412124
Title: Quality of Life Outcomes From a Peer-to-Peer Support Program for Women With Gynecologic Cancer
Brief Title: Peer-to-Peer Support Program in Improving Quality of Life Outcomes in Patients With Gynecologic Cancer and Their Caregivers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility issues
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14359; NCI-2015-00467 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14359 (Other: City of Hope Medical Center)
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Cervical Carcinoma; Ovarian Carcinoma; Uterine Corpus Cancer; Vaginal Carcinoma; Vulvar Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (W2W program) (Experimental): Patients participate in the W2W program for which they are matched with a trained mentor and followed throughout treatment by phone, email, and/or in person.
  Interventions: Procedure: Supportive Care; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Supportive Care — Complete W2W mentoring program
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
Other: Quality-of-Life Assessment — Complete the FACT-G
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete the W2W Patient Survey

SUMMARY:
This pilot clinical trial studies a peer-to-peer support program in improving quality of life outcomes in patients with gynecologic cancer and their caregivers. Peer-to-peer support and mentoring may help improve quality of life and reduce symptoms of distress in gynecologic cancer patients and their families.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the feasibility and acceptability of a Woman-to-Woman (W2W) program for patients with gynecologic cancer at City of Hope (COH). Address the following descriptive research questions: were patients, mentors, and patients' family caregivers satisfied with the timing, format, and content of the program? Did the program benefit patients, mentors, and patients' family caregivers?

OUTLINE:

Patients participate in the W2W program for which they are matched with a trained mentor and followed throughout treatment by phone, email, and/or in person.

After completion of study, patients are followed up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT PARTICIPANTS
* Patients with newly diagnosed or recurrent gynecologic cancer (ovarian, uterine, cervical, vaginal, vulvar) actively undergoing treatment (chemotherapy, surgery, or radiation therapy) at COH (including Duarte and South Pasadena campuses)
* English-speaking patients
* PEER MENTORS
* Peer mentors will be past gynecologic cancer patients not currently undergoing treatment for their cancer, and considered without evidence of disease
* Over age 18
* PEER MENTORS: English-speaking patients
* This study is open to patients of all races and ethnicities

Exclusion Criteria:

* PEER MENTORS:
* Major psychiatric disease
* Currently undergoing treatment for active gynecologic cancer

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-07; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in quality of life benefits for patients, as assessed by the FACT-G | Baseline to up to 12 months
  Changes from baseline will be tested using paired t-tests. Data will be summarized using descriptive statistics, including means for normally distributed continuous data, medians for non-normally distributed continuous data or proportions for categorical data. Established instruments will be scored according to standard instructions, and appropriate descriptive statistics computed. Written comments from all open ended questions analyzed using content analysis methods.
Satisfaction of patients with the timing, content, and format of the program, as assessed by the W2W Patient Survey | Up to 12 months
  Changes from baseline will be tested using paired t-tests. Descriptive statistics on participants' satisfaction with the timing, content, and format of the intervention will be presented through summary statistics of data from the satisfaction tools. Data will be summarized using descriptive statistics, including means for normally distributed continuous data, medians for non-normally distributed continuous data or proportions for categorical data.
Satisfaction of mentors with the timing, content, and format of the program, as assessed by the W2W Volunteer/Mentor Survey | Up to 12 months
  Descriptive statistics on participants' satisfaction with the timing, content, and format of the intervention will be presented through summary statistics of data from the satisfaction tools.
Satisfaction of patients' family caregivers with the timing, content, and format of the program | Up to 12 months
  Changes from baseline will be tested using paired t-tests. Descriptive statistics on participants' satisfaction with the timing, content, and format of the intervention will be presented through summary statistics of data from the satisfaction tools.
Benefits for patients' family caregivers after participating in the program, as assessed by the Modified Caregiver Strain Index | Up to 12 months
  Data will be summarized using descriptive statistics, including means for normally distributed continuous data, medians for non-normally distributed continuous data or proportions for categorical data. Established instruments will be scored according to standard instructions, and appropriate descriptive statistics computed. Written comments from all open ended questions analyzed using content analysis methods.

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Dellinger, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States